CLINICAL TRIAL: NCT07153549
Title: A Parallel-Group, Randomized, Open-Label, Controlled Study to Evaluate the Efficacy and Safety of a Zinc-Containing Dietary Supplement (Biolizin) in Improving Functional Poor Appetite in Children Aged 6 to 36 Months
Brief Title: Biolizin for Improving Functional Poor Appetite in Children Aged 6 to 36 Months (CTBE2502)
Acronym: CTBE2502
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTBE.25.02; Protocol No.: CTBE.25.02 (Other: Clinical Trial and Bioequivalence Center - Hai Phong University of Medicine and Pharmacy)
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Feeding and Eating Disorders of Childhood; Appetite Disorders; Functional Poor Appetite
Keywords: functional poor appetite; pediatric feeding problems; feeding difficulty; loss of appetite; eating/feeding behavior; Children's Eating Behaviour Questionnaire; toddler; infants; zinc supplement; dietary supplement; Biolizin
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Feeding and Eating Disorders; Anorexia; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Two groups: zinc-containing oral supplement (Biolizin) plus standardized caregiver counseling versus counseling only; follow-up for 42 days; age-stratified randomization (6-12 vs 13-36 months)
Masking Description: Not applicable (open-label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biolizin Syrup + Standardized Caregiver Counseling (Experimental): Children receive an oral zinc-containing dietary supplement (Biolizin syrup) for 42 days, dosed by age per protocol, together with standardized caregiver counseling on responsive feeding at each study visit (Day 0, Day 7, Day 21, Day 42). Adherence is monitored with dosing diaries and returned bottle counts. Use of other zinc-containing products or appetite stimulants is not permitted. Outcomes (feeding-difficulty score, CEBQ subscales, anthropometrics, and safety labs) are collected per schedule
  Interventions: Dietary Supplement: Biolizin; Behavioral: Standardized caregiver counseling on responsive feeding
- Counseling Only (Standardized Feeding-Behavior Counseling) (Active Comparator): Children receive the same standardized caregiver counseling on responsive feeding at each study visit (Day 0, Day 7, Day 21, Day 42) without Biolizin or any other zinc-containing supplement. Education materials, visit frequency, and assessments match the experimental arm. Concomitant appetite stimulants or zinc products are not allowed. Outcomes are collected per the same schedule.
  Interventions: Behavioral: Standardized caregiver counseling on responsive feeding

INTERVENTIONS:
Dietary Supplement: Biolizin — Oral zinc-containing syrup taken per age-based dosing specified in the protocol, once or twice daily for 42 consecutive days. Product is dispensed at baseline (with refill if needed); batch and expiry are recorded. Caregivers receive instructions for use and complete dosing diaries; adherence is checked by diary review and returned bottle counts. Concomitant zinc products or pharmacologic appetite stimulants are not allowed. Safety is monitored through adverse event review and routine laboratory tests at baseline and Day 42.
  Arms: Biolizin Syrup + Standardized Caregiver Counseling
Behavioral: Standardized caregiver counseling on responsive feeding — Structured counseling delivered to caregivers at each clinic visit (Day 0, Day 7, Day 21, Day 42). Content includes mealtime routines, recognizing hunger/satiety cues, age-appropriate portions and textures, repeated exposure to diverse foods, and strategies to manage refusal or prolonged meals. A brief checklist guides delivery to ensure consistency across visits. No dietary supplement is provided in this intervention.

SUMMARY:
Functional poor appetite is common in young children and may be linked to suboptimal micronutrient intake and feeding behavior. This study evaluates whether a zinc-containing oral supplement (Biolizin syrup) can improve eating behavior in children aged 6 to 36 months who have poor appetite without an identifiable medical cause. Participants are followed for 42 days with clinic visits at Day 0, Day 7, Day 21, and Day 42. Caregivers complete validated questionnaires about feeding difficulties and eating behavior; the child's weight and length/height are measured at each visit. Safety is assessed through review of adverse events and routine laboratory tests; serum zinc may be measured according to the protocol. The primary outcome is the change from baseline to Day 42 in the total score of a validated feeding-difficulty scale. Secondary outcomes include changes in Children's Eating Behaviour Questionnaire (CEBQ) subscales, WHO growth indices, serum zinc (if measured), and overall safety

DETAILED DESCRIPTION:
Poor appetite in toddlers often reflects a combination of nutritional and behavioral factors. Zinc is an essential trace element that contributes to taste perception, mucosal integrity, and appetite regulation; suboptimal zinc status may exacerbate reduced intake and feeding problems. Biolizin is an oral zinc-containing supplement intended to support appetite and healthy feeding behavior in young children. The study aims to determine whether the supplement, provided together with standardized caregiver counseling on responsive feeding practices, improves caregiver-reported feeding difficulty and eating behavior over 42 days. After consent and screening, eligible children attend visits at Day 0, Day 7 (±2), Day 21 (±3), and Day 42 (±4). At each visit, clinicians review medical history and concomitant treatments, record anthropometrics, and caregivers complete a validated Vietnamese feeding-difficulty scale (0-24, higher scores indicate worse difficulty) and the CEBQ subscales. The study product is taken orally per age-based dosing specified in the protocol; adherence is checked using dosing diaries and returned bottle counts where applicable. Safety laboratories (e.g., complete blood count, liver and renal chemistry) are planned at baseline and Day 42; serum zinc may be obtained according to protocol. Adverse events are collected from consent through Day 42 and are managed according to clinical judgment; expected reactions are generally mild (for example, gastrointestinal discomfort, taste changes, or rash). Source data are recorded in case report forms and entered into a secure database with audit trails, and only de-identified data are used for analysis or sharing. The study has ethics approval and written informed consent is obtained from caregivers before any procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 36 months at screening.
* Functional poor appetite for ≥2 weeks with at least one of the following:

  * Clearly reduced intake versus usual (lower amount of food and/or fewer meals per day);
  * Prolonged meal duration (>30 minutes per meal);
  * Refusal or avoidance of familiar foods previously accepted;
  * Oppositional feeding behaviors (turning away, crying, gagging/retching, prolonged food holding, lack of cooperation during meals).
* No obvious organic cause of poor appetite (e.g., acute infection, gastrointestinal/metabolic disease).
* Weight not below -2 SD compared with WHO growth standards.
* Parent/guardian provides written informed consent.

Exclusion Criteria:

* Ongoing acute or chronic illnesses that can affect intake or absorption, including but not limited to:

  * Acute infections (e.g., tonsillitis, pneumonia, otitis media, viral febrile illness, acute diarrhea);
  * Chronic conditions affecting digestion or metabolism (e.g., celiac disease, malabsorption syndromes, chronic liver disease, chronic kidney disease, diabetes).
* Neurodevelopmental or neurological conditions that impair feeding (e.g., cerebral palsy, autism spectrum disorder, global developmental delay).
* Current or recent use of medications known to alter appetite or digestion/absorption (e.g., systemic corticosteroids, antiepileptics, prolonged antibiotics).
* Use of zinc-containing products or other appetite stimulants within 7 days before screening.
* Known hypersensitivity to any component of the study product.
* Malabsorption, severe malnutrition, or requirement for specialized nutrition, including:

  * Confirmed or suspected malabsorption (e.g., celiac disease, severe lactose intolerance, short bowel syndrome, inflammatory bowel disease);
  * Severe malnutrition per WHO criteria (e.g., weight-for-length Z-score < -3 SD, nutritional edema, marked loss of subcutaneous fat/muscle);
  * Physician-prescribed specialized nutrition plans (therapeutic formulas for cow's milk protein allergy, severe malnutrition, tube feeding, or individualized nutrition regimens beyond usual diet).
* Nonadherent caregiver or high risk of loss to follow-up as judged by the investigator.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Eating Behaviour Questionnaire (CEBQ) Composite Total Score from Baseline to Day 42 | Baseline to Day 42
  The CEBQ is a validated parent-reported questionnaire assessing eating behaviors in children. Each item is scored from 1 (never) to 5 (always). The composite total score is derived from multiple domains (range: 1-5). Higher scores indicate more adverse eating behaviors (worse outcome). A negative change (Day 42 - Baseline < 0) indicates improvement.
Change in Children's Eating Behaviour Questionnaire (CEBQ) Food Approach Behaviors from Baseline to Day 42 | Baseline to Day 42
  The Children's Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported questionnaire assessing eating behaviors in children. The "food approach" score is the mean of four subscales: Enjoyment of Food, Food Responsiveness, Emotional Overeating, and Desire to Drink. Each item is scored from 1 (never) to 5 (always). Subscale scores range from 1-5, with higher values indicating greater food approach behaviors (worse outcome). A negative change indicates improvement.
Change in Children's Eating Behaviour Questionnaire (CEBQ) Food Avoidant Behaviors from Baseline to Day 42 | Baseline to Day 42
  Mean change in Children's Eating Behaviour Questionnaire (CEBQ) "food avoidant" subscales (Satiety Responsiveness, Slowness in Eating, Food Fussiness, Emotional Undereating). Lower scores indicate less avoidance; negative change denotes improvement.
Responder Rate on Children's Eating Behaviour Questionnaire (CEBQ) (≥30% Improvement) at Day 42 | Day 42
  Proportion of participants achieving ≥30% decrease from baseline in the pre-specified Children's Eating Behaviour Questionnaire (CEBQ) adverse-behavior composite (per SAP).

SECONDARY OUTCOMES:
Change in Hoang Thi Bach Yen Anorexia Scale (Vietnamese Caregiver-Reported Pediatric Anorexia Scale) Total Score from Baseline to Day 42 | Baseline to Day 42
  The Hoang Thi Bach Yen Anorexia Scale (2020) is a validated Vietnamese caregiver-reported instrument to assess poor appetite in children. It includes 8 items covering mealtime characteristics (duration, amount of food intake) and eating behaviors (oppositional behavior, avoidance, food selectivity, food refusal). Each item is scored from 0 to 3 (0 = no symptom, 3 = severe symptom). The total score ranges from 0 to 24. Higher scores indicate worse appetite (more severe anorexia). Lower scores indicate better appetite. A negative change (Day 42 - Baseline < 0) reflects clinical improvement.
Change in Body Weight from Baseline to Day 42 | Baseline to Day 42
  Body weight will be measured in kilograms (kg) at baseline and Day 42. The outcome is the mean change (Day 42 - Baseline). Weight-for-age Z-scores based on WHO growth standards may also be summarized descriptively.
Change in Number of Daily Meals from Baseline to Day 42 | Baseline to Day 42
  Caregiver-reported average number of meals per day over the prior week; outcome is change (Day 42 - Baseline).
Change in Mean Meal Duration from Baseline to Day 42 | Baseline to Day 42
  Caregiver-reported average minutes per meal over the prior week; outcome is change (Day 42 - Baseline).
Change in Caregiver-Rated Cooperation During Meals Scale Score from Baseline to Day 42 | Baseline to Day 42
  Caregiver-Rated Cooperation During Meals Scale is a study-specific, caregiver-reported measure of mealtime cooperation. The instrument uses a 5-point Likert scale ranging from 1 (very uncooperative) to 5 (very cooperative). Higher scores indicate better cooperation (favorable outcome). A positive change (Day 42 - Baseline > 0) reflects improvement.
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) | From first dose to Day 42
  Number and proportion of participants with ≥1 TEAE; events characterized by system organ class/preferred term and graded by CTCAE v5.0. Collected using the study's standard ADR form.
Change in Serum Zinc Concentration from Baseline to Day 42 | Baseline to Day 42
  Serum zinc (µg/dL) measured per site laboratory procedures; outcome is change (Day 42 - Baseline).
Change in Body Length/Height from Baseline to Day 42 | Baseline to Day 42
  Body length (for children <24 months) or standing height (for children ≥24 months) will be measured in centimeters (cm) at baseline and Day 42. The outcome is the mean change (Day 42 - Baseline). Length/height-for-age Z-scores based on WHO growth standards may also be summarized descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial and Bioequivalence Center, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcomes will be shared, including: baseline demographics/clinical characteristics; CEBQ item- and subscale-level scores and the prespecified composite; Hoang Thi Bach Yen anorexia scale scores; anthropometrics and WHO Z-scores; serum zinc and laboratory safety values; adverse events; concomitant medications; intervention assignment and adherence. A data dictionary/codebook will accompany the dataset. Direct identifiers will be removed and indirect identifiers minimized per protocol and institutional policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will be available beginning ~6-12 months after publication of the primary results and for 36 months thereafter. If no publication occurs, availability will begin within 24 months after last patient last visit and continue for 36 months.
Access Criteria: Qualified researchers from academic, non-profit, or health-care institutions may request access by submitting a methodologically sound proposal and analysis plan to the Sponsor/PI (see Contacts). Requests require IRB/ethics determination or waiver and a signed Data Use Agreement. Upon approval, de-identified data and documents will be provided via secure, access-controlled repository or encrypted file transfer. Re-identification attempts and onward sharing are prohibited; use is limited to the approved objectives.